CLINICAL TRIAL: NCT01419418
Title: A Study of Patients' Perspectives of Factors That Support the Management of Cardiac Care for Improved Outcomes in a Peripheral Arterial Disease Population
Brief Title: Patients' Perspectives of Factors That Support the Management of Peripheral Arterial Disease for Improved Outcomes
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anne Lambert-Kerzner, Health Services Researcher, VA Eastern Colorado Health Care System
Other Study IDs: 10-1361
Record Dates: First submitted 2011-04-11; First posted 2011-08-18 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Peripheral Arterial Diseases
Keywords: Peripheral Arterial Disease (PAD); Qualitative analysis; Patients' perspective
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peripheral Arterial Disease (PAD): This is a longitudinal observational study. There were no interventions administered.

SUMMARY:
Specific Aims: To delve into the complex phenomena of living with Peripheral Arterial Disease (PAD), and to investigate the patients' perspective of the factors that affects their decisions regarding management of their PAD.

a) Utilize a qualitative approach to uncover factors that patients perceive support the management of their condition utilizing a purposive sampling of Peripheral Arterial Disease patients.

1. To determine what they believe to be effective tools to support themselves to improve their condition.
2. To determine from the patient's perspective if adherence to prescribed medical regimes are important for them to improve their PAD outcomes.
3. To describe the patient factors of those who are self reported adherent compared to those who are not or unable to their prescribed regimen.

DETAILED DESCRIPTION:
Cardiovascular Diseases (CVD) affects as many lives each year as cancer, chronic lower respiratory diseases, accidents and diabetes mellitus combined. One in three American adults (about 80,000,000) has one or more types of cardiovascular disease. Prevention and management of CVD is a public health goal, yet, it remains a major challenge. Even hypertension, which is easily detected and usually controllable, has only a 50 percent control rate.

Peripheral Arterial Disease (PAD) is one type of CVD, which affects about eight million Americans and is also associated with significant morbidity and mortality. PAD increases with age and disproportionately affects African Americans. Interestingly, despite its prevalence and cardiovascular risk implications, only 20 to 30 percent of PAD patients are undergoing treatment.

Medical management of these diseases has substantially contributed to improved morbidity and mortality. However, for the medical therapies to be successful the patients need to take their medications and adjust their lifestyles, as prescribed. Overall, "typical adherence rates for the general population are about 50 percent for medications and are much lower for lifestyle prescriptions and other more behaviorally demanding regimens". Few studies have investigated the reactions and thoughts regarding the efficacy of therapies/interventions from the perspective of the participants. Meta analyses on adherence have also revealed that the patients' perspectives are often absent and that present adherence theories are more successful in explaining non-adherence than improving adherence. Therefore, it is important to understand, from the perspective of the patient; the factors they believe improve their cardiac outcomes with an emphasis on the adherence to prescribed therapies.

This qualitative study will investigate the question: What are patients' perspectives of factors that support the management of their cardiovascular condition to improve outcomes in a Peripheral Arterial Disease population? Cardiac outcomes of interest are health status defined by symptom burden, functional status, and health related quality of life, patients' perception of the quality of care that they receive, and the experience of living with PAD.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Peripheral Arterial Disease

Exclusion Criteria:

Unable to converse about the topic under investigation for up to one hour for multiple visits

Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A purposive sampling technique, meaning the sample will be selected according to the participant's diagnosis of the specific disease, will be utilized to enroll up to 24 Peripheral Arterial Disease patients from the VA Peripheral Arterial Disease clinic.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patients' perspective of the factors that affects their decisions regarding management of their PAD | 1 year
  Qualitative interview that will collect patients perspectives and will be analyzed for thoughts, opinions, feelings, and concepts.

SECONDARY OUTCOMES:
Quantitative Morinsky's Medication adherence survey | 1 year
  Morinsky's Medication adherence survey will be administered at baseline and one year to assess self report medication adherence.
Quantitative PAQ health status survey | 1 year
  PAQ health status will be administered at the initial visit as well as the last one-on-one interview to assess disease specific health status.
Quantitative EQ-5D health status survey | 1 year
  survey will be administered at the initial visit as well as the last one-on-one interview to assess overall health status.
Quantitative Stage of Change Survey | 1 year
  Stage of Change motivational survey will be administered at the initial visit as well as the last one-on-one interview to assess patients motivational status.
Quantitative SEAMS survey | 1 year
  SEAMS self efficacy survey will be administered at the initial visit as well as the last one-on-one interview to assess patient self efficacy to adhere to medication treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Lambert-Kerzner, PhD, MSPH, Principal Investigator — VAMC in Denver, Co.; Thomas Tsai, MD, Study Director — VAMC Denver, Co.
Locations (1):
- VA ECHCS, Denver, Colorado, United States